CLINICAL TRIAL: NCT03174951
Title: Effect of IVIg on Pregnancy Rate of Patient With Recurrent Pregnancy Loss With Immunological Causes
Brief Title: Immunomodulatory Effects of IVIg on Pregnancy Rate of Patient With Recurrent Pregnancy Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TabrizUMS-infertility-003
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Recurrent Pregnancy Loss; IVIg; Pregnancy Rate
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): IVIg group
  Interventions: Drug: IVIg
- control group (No Intervention): Patients who do not receive any treatment despite a history of Recurrent Pregnancy Loss problem as controls

INTERVENTIONS:
Drug: IVIg — Patients will take 400mg/kg IVIg at the time of positive pregnancy,Following the first administration, IVIG well given every 4 weeks through 32 weeks of gestation.
  Arms: Treatment group

SUMMARY:
Miscarriage occurs in about 1-2% of human pregnancies and is one of the common pregnancy problems before 12 weeks of pregnancy. Anatomical and chromosomal abnormalities, microbial factors and auto and alloimmune reactions have been speculated to attribute in recurrent miscarriage. Unexplained recurrent miscarriage (URM) is defined as three or more repeated abortions, probably caused by maternal immunological rejection . Given that maternal immune system encounters semi-allogeneic fetus, pregnancy outcome is associated with the interaction between maternal immune system and immuno-regulatory capability of the fetus. Effectiveness of treatment approaches in RM patients has been controversial and remained to be discovered. Immunomodulatory agents such as corticosteroids and allogeneic lymphocyte immunization showed variable success rates in RM patients. Therapeutic effects of IVIG in unexplained RM is controversial and most positive results were obtained from the trials in RM women with cellular immune abnormalities, such as increased NK cell level and/or cytotoxicity, and T cell abnormalities. Previous studies have shown that the incidence of genetic abnormalities in children who have received immunosuppressive drugs such as IVIg like normal people and normal society. In this study we used IVIg at the time of positive pregnancy,400 mg/kg IVIG was administered intravenously. Following the first administration, IVIG well given every 4 weeks through 32 weeks of gestation to suppress the immune system in patients with immunological causes of RPL and the results will be compared with a control group that did not receive any type of drug.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients will experience at least 3 times recurrent pregnancy loss.
* Patients dont have history of any type of immunotherapy.
* Patients must have abnormal NK cell or NK cell cytotoxicity or Th1/Th2 ratio

Exclusion Criteria:

- Our criteria for exclusion of patients from the study include the following:

* Patients or their spouse has abnormal karyotype or chromosomal and genetically disorders.
* Patients who have bleeding problems.
* Patients who have chronic disorders those are forced to use the specific drug.
* Patients who have positive test for HIV, HCV or HBV infection.
* Patients who have a history of asthma and allergies.
* Patients who have uterus abnormalities.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in NK cells, T reg and Th17 cells frequency. | up to 8 month of pregnancy
  Flowcytometry
Changes in secretion levels of cytokines related to Treg and Th17 cells(IL-17,IL-21) | up to 8 month of pregnancy
  Elisa
Changes in exoression of cytokines gene. | up to 8 month of pregnancy
  RT pcr

SECONDARY OUTCOMES:
Ongoing pregnancy rate in patients with Recurrent Pregnancy Loss (RPL) | up to 8 month of pregnancy
  by sonography
Live berth rate in patients with Recurrent Pregnancy Loss (RPL). | up to 1 year
  Monitoring by gynecologists

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nouri, Ph.D, Study Chair — Head of SCARM institute; Mehdi Yousefi, Immunologist, Study Director — SCARM institute
Locations (1):
- Alzahra hospital, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sugiura-Ogasawara M, Suzuki S, Ozaki Y, Katano K, Suzumori N, Kitaori T. Frequency of recurrent spontaneous abortion and its influence on further marital relationship and illness: the Okazaki Cohort Study in Japan. J Obstet Gynaecol Res. 2013 Jan;39(1):126-31. doi: 10.1111/j.1447-0756.2012.01973.x. Epub 2012 Aug 13. PMID 22889462
- [Result] Santos MA, Kuijk EW, Macklon NS. The impact of ovarian stimulation for IVF on the developing embryo. Reproduction. 2010 Jan;139(1):23-34. doi: 10.1530/REP-09-0187. PMID 19710204
- [Result] King K, Smith S, Chapman M, Sacks G. Detailed analysis of peripheral blood natural killer (NK) cells in women with recurrent miscarriage. Hum Reprod. 2010 Jan;25(1):52-8. doi: 10.1093/humrep/dep349. Epub 2009 Oct 9. PMID 19819893
- [Result] Goring SM, Levy AR, Ghement I, Kalsekar A, Eyawo O, L'Italien GJ, Kasiske B. A network meta-analysis of the efficacy of belatacept, cyclosporine and tacrolimus for immunosuppression therapy in adult renal transplant recipients. Curr Med Res Opin. 2014 Aug;30(8):1473-87. doi: 10.1185/03007995.2014.898140. Epub 2014 Apr 3. PMID 24628478
- [Result] Yamada H, Morikawa M, Furuta I, Kato EH, Shimada S, Iwabuchi K, Minakami H. Intravenous immunoglobulin treatment in women with recurrent abortions: increased cytokine levels and reduced Th1/Th2 lymphocyte ratio in peripheral blood. Am J Reprod Immunol. 2003 Feb;49(2):84-9. doi: 10.1034/j.1600-0897.2003.01184.x. PMID 12765346
- [Result] Hutton B, Sharma R, Fergusson D, Tinmouth A, Hebert P, Jamieson J, Walker M. Use of intravenous immunoglobulin for treatment of recurrent miscarriage: a systematic review. BJOG. 2007 Feb;114(2):134-42. doi: 10.1111/j.1471-0528.2006.01201.x. Epub 2006 Dec 12. PMID 17166218
- [Result] Kolls JK, Khader SA. The role of Th17 cytokines in primary mucosal immunity. Cytokine Growth Factor Rev. 2010 Dec;21(6):443-8. doi: 10.1016/j.cytogfr.2010.11.002. Epub 2010 Nov 20. PMID 21095154